CLINICAL TRIAL: NCT06963970
Title: Using Community Health Workers to Support Rural Care Partners of Seriously Ill Older Veterans
Acronym: PATH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SDR 24-078; 1l01HX003922-01A1 (Other Grant/Funding Number: Veterans Administration)
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Dementia; Cancer; Renal Disease; Obstructive Pulmonary Disease
MeSH Terms: conditions — Dementia; Neoplasms; Kidney Diseases; Lung Diseases, Obstructive

STUDY DESIGN:
Intervention Model Description: Enrolled Care Partners are randomized to the study. The control arm is care partners of seriously ill veterans who are enrolled in the Caregiver Support Program and the intervention arm is care partners of seriously ill veterans who are enrolled in the Caregiver Support Program PLUS receiving a study-provided community health worker for additional support.
Who Masked: Outcomes Assessor
Masking Description: Study staff collecting baseline and 6 month measures will be masked to the arm enrollment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community Health Worker support (Experimental): Additional weekly remote support of care partner using a trained/certified community health worker
  Interventions: Other: Remote Community Health Worker support
- Regular support (No Intervention): Regular care

INTERVENTIONS:
Other: Remote Community Health Worker support — trained/certified community health worker supporting care partner remotely
  Arms: Community Health Worker support

SUMMARY:
The investigators aim to support care partner's well-being and satisfaction with VA care and decrease their work burden by offering extra support from a trained Community Health Worker who will help connect the care partner to helpful resources in their communities and in the VA. The investigators also hope to help Veterans well-being and satisfaction with VA care by supporting their care partner more sufficiently allowing the care partner to focus on caregiving tasks.

DETAILED DESCRIPTION:
Aim 1: Determine CSNAV effectiveness in increasing rural Veterans' well-being, reducing rural care partner burden, and increasing rural care partner/Veteran satisfaction with VA care in the intervention group compared with the usual care (CSP) group. The investigators will apply a 6-month intervention in a randomized control trial over 27 months. Primary Outcome: (H1) Care partners randomized to intervention group will have lower mean Zarit-1216 burden scores at 6 months compared to the control group. Secondary Outcomes: (H2) Care partners and Veterans randomized to the intervention group will have higher mean CAHPS Global Satisfaction17 scores at 6 months compared to the control group. (H3) Veterans randomized to the intervention group will have higher mean Warwick Edinburgh Mental Well-Being Scale18 scores at 6 months compared to the control group.

Aim 2: Following intervention, the investigators explore Veterans' and care partners' experience of CHWs as a mode of VA support using semi-structured interviews. The investigators then facilitate Delphi Method sessions with the Community Advisory Board plus study Veterans/care partners, CHWs, and key operational partners to examine Aims 1 & 2 data for intervention improvements and implementation planning using updated CFIR.19

Aim 3: Conduct budget impact analysis from the VA perspective to evaluate cost-drivers and assess feasibility to inform adaptation and implementation of the intervention within a VA regional network.

ELIGIBILITY:
Inclusion Criteria:

Care Partner Inclusion Criteria

* A relative, friend, or partner (18 years of age) with whom Veteran patient has a personal relationship who assists Veteran regularly with care and/or care coordination as defined under "Veterans" below
* Residing in a rural area based on RUCC or Rural-Urban Continuum Codes83
* Must be enrolled in CSP Program of General Caregiver Support Services
* Can live with or separately from the Veteran; able to communicate in English by phone

Veteran Inclusion Criteria

* Receiving care at Durham, Asheville, and Richmond VA Health Systems (e.g., at least 2 outpatient visits in past year; has a primary provider) and residing in a rural area.
* Diagnosed with congestive heart failure, chronic obstructive pulmonary disease, cancer, dementia, or end-stage renal disease.
* Requires assistance with at least one ADL (i.e., walking, feeding, toileting, transferring, bathing, or dressing) or IADL (i.e., transport, medication, financial management, shopping, or meal preparation)
* 50 years old or older and able to communicate in English by phone (for assessments)

Exclusion Criteria:

Veteran Exclusion Criteria

* Flag or social work note indicating suspected Caregiver abuse.
* Unable to communicate in English by phone for assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Zarit-12 Cargiver Burden Interview | baseline and 6 months
  Care partners randomized to intervention will have lower mean Zarit-12 scores at 6 months compared to the control group. Each question is scored on a five-point Likert scale from 0 to 4, with higher scores representing a greater feeling of burden. The total ZBI-12 score is the summation of 12 items, with a total score range from 0 to 484. Higher indicates more burden.
  A cut-off score of 13 points on the ZBI-12 is suggested for screening burden in community-dwelling older caregivers, but should not be assumed as normative data.
  5 categories: health, psychological well-being, finances, social life, relationship with impaired person. 12 item, α=0.88-0.91

SECONDARY OUTCOMES:
1-item CAHPS Global Satisfaction Measure | baseline and 6 months
  Care partners and Veterans randomized to intervention will have higher mean 1-item CAHPS Global Satisfaction scores at 6 months compared to the control group. Scale of 0 to 10 to measure respondents' overall assessments of a provider, care, and/or healthcare organization. Higher score means a more satisfied.
Warwick Edinburgh Mental Well-Being Scale | baseline and 6 months
  Veterans randomized to intervention will have higher mean Warwick Edinburgh Mental Well-Being Scale scores at 6 months compared to the control group. 14 item scale (scored 1-5) of mental well-being covering subjective well-being and psychological functioning, in which all items are worded positively and address aspects of positive mental health. The minimum scale score is 14 and the maximum is 70, higher is more positive well-being. α=0.89-0.91
Connection Measure | baseline and 6 months
  1. At baseline and 6 months. "When I need services at the VA, I was connected to those services" Strongly Agree-Agree-Disagree-Strongly Disagree Scale
     o At 6 months only: In what ways has connecting to services at VA changed for you since the beginning of the study? Open-ended response
  2. At baseline and 6 months. "When I need services in my community, I was connected to those services" Strongly Agree-Agree-Disagree-Strongly Disagree Scale
     * At 6 months only: In what ways has connecting to services in the community changed for you since the beginning of the study? Open-ended response

CONTACTS AND LOCATIONS:
Overall Officials: Nathan A Boucher, DrPH, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No